CLINICAL TRIAL: NCT00858923
Title: Phase 1 Study of the HemoModulator System for the Treatment of Human Immunodeficiency Virus (HIV)
Brief Title: Safety Study of the HemoModulator System for the Treatment of Patients With Human Immunodeficiency Virus (HIV)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Energex Systems, Inc. (Industry)
Responsible Party: David M. Mushatt, MD, Tulane U. Health Sciences Center/Louisiana Community AIDS Research Program
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G080104
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-03

CONDITIONS: HIV; HIV Infections
Keywords: Extracorporeal Photophoresis; immuno-therapy; treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Energex HemoModulator — To use ultraviolet light to reduce HIV virus in the patient's blood
  Other Names: Extracorporeal photophoresis

SUMMARY:
Tulane University Health Sciences Center/Louisiana Community AIDS Research

Center Program, New Orleans, LA is seeking patients for an HIV study. The

purpose of the study is to test the safety and effectiveness of an

experimental ultra-violet light device designed to reduce virus in your blood.

DETAILED DESCRIPTION:
You may be eligible if:

* You have HIV
* Your CD4 cell count is or greater than 400
* Your viral load is greater than 10,00 copies
* You do not yet qualify for standard antiviral therapy (HAART)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV-1 has been confirmed positive by ELISA and by Western Blot
* Subject is not yet eligible for HAART
* Subject's viral count at pre-baseline measured by RT-PCR is

  * 10,000 copies /ml
* Subject has a CD4+ count ≥ 400 cells/mm3
* Subject's pre-screen EIA and RIBA test has proven negative for Hepatitis C virus
* Female subjects with reproductive potential (and any male sexual partners) must agree to use a barrier device with spermicide (e.g., condoms, cervical cap, diaphragm) as the primary form of contraception, in addition to any other methods used, during treatment and until the end of the study to prevent pregnancy
* Subject has taken no other anti-viral device or pharmacologic treatments in the 2 months prior to the first scheduled Hemo-Modulator study treatment
* Subject agrees not to receive any other anti-viral device or anti-viral pharmacologic treatment (including herbal remedies) throughout the 21-week study period
* Subject weighs at least 90 lbs (40.9 kg) at study initiation
* Subject agrees to comply with study protocol requirements including all follow up visits through Day 60 of study duration

Exclusion Criteria:

* Subjects with any other major illness (e.g., malignancy, renal failure, tuberculosis, porphyria, severe cardiac disease, severe neurological disease, or Hepatitis C) that would prevent completion of the study or bias efficacy assessments
* Subjects with any other medical condition that the Investigator believes would make the patient unable to safely tolerate the extracorporeal blood volume required during the procedure [e.g., severe cardiovascular disease, history of congestive heart failure, or severe anemia (hemoglobin < 90 g/L)]
* Subject with porphyria cutanea tarda (PCT), since PCT is associated with increased sensitivity to light and skin reactions such redness, pain, swelling and blistering after exposure to ultraviolet light
* Subject has clinically abnormal hemotologic or chemistry laboratory values, defined as any parameter for these tests that exceeds Grade 1 (DAIDS Table for Grading the Severity of Adult Adverse Events, December 2004)
* Subject has taken a steroid drug (other than Estrogen or Progesterone) within 7 days prior to study enrollment, or may require such medications during the course of study participation
* Subject has taken a drug listed as photosensitizing in the Physician's Desk Reference (PDR) within 7 days prior to a Hemo-Modulator Treatment session
* Subjects that habitually use excessive alcohol
* Subjects that use illicit drugs or have an ongoing drug abuse problem
* Subjects that have an acute systemic bacterial infection (septicemia)
* Subjects that have been immunized for influenza within 7 days prior to study enrollment or is likely to require such immunization during the course of study participation
* Subject is currently participating in another clinical investigation of a medical device, drug or biologic, or has participated in such a study within the 3 months prior to study enrollment
* Subject is pregnant or plans on becoming pregnant within the next twelve months; or is lactating
* Subject has a clotting deficiency
* Subject is allergic to heparin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Determine the therapy effectiveness on HIV-1 plasma viral load using PCR analysis Determine the therapy effects on CD4+, CD8+ cells and CD4/CD8 ratio | Once a week for 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane University Health Sciences Center/LaCarp, New Orleans, Louisiana, United States